CLINICAL TRIAL: NCT06844383
Title: A Randomized Open-label Phase 2 Study of TALazoparib With or Without ENzaluTamide in Patients With Metastatic Castration-Resistant Prostate Cancer and HRR Mutations After Progression on Abiraterone Acetate
Brief Title: A Study of Talazoparib With or Without Enzalutamide in People With Prostate Cancer Who Have Previously Received Abiraterone Acetate
Acronym: TALENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prostate Cancer Clinical Trials Consortium (Other)
Collaborators: Pfizer (Industry); Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: c24-349
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer (Adenocarcinoma); mCRPC (Metastatic Castration-resistant Prostate Cancer)
Keywords: talazoparib; enzalutamide; PARP inhibitor; TALENT; androgen receptor signaling inhibitor (ARSI); Prostate Cancer Clinical Trials Consortium, LLC (PCCTC); c24-349
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — talazoparib; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Talazoparib (0.5 mg PO QD) and enzalutamide (160 mg PO QD) will be administered in continuous 28-day cycles.
  Interventions: Drug: Talazoparib with enzalutamide
- Arm B (Experimental): Talazoparib (1 mg PO QD) will be administered in continuous 28-day cycles.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib with enzalutamide — Talazoparib (0.5 mg PO QD) and enzalutamide (160 mg PO QD) will be administered in continuous 28-day cycles.
  Other Names: Talzenna; Xtandi
  Arms: Arm A
Drug: Talazoparib — Talazoparib (1 mg PO QD) will be administered in continuous 28-day cycles.
  Other Names: Talzenna
  Arms: Arm B

SUMMARY:
The purpose of this study is to find out whether talazoparib in combination with enzalutamide or talazoparib alone delays cancer progression in people with metastatic castration-resistant prostate cancer (mCRPC) who have homologous recombination repair (HRR) mutations and have previously received abiraterone acetate.

ELIGIBILITY:
Inclusion Criteria

• Willing and able to provide, or have a legally authorized representative provide, written informed consent and privacy authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.

NOTE: Privacy authorization may be either included in the informed consent or obtained separately.

* Participants ≥ 18 years of age.
* Are willing to be randomized into either study arm and adhere to the study protocol.
* Ability to swallow study capsules and/or tablets whole.
* Are willing to remain on study treatment and to continue undergoing study imaging despite PSA progression unless clinically deteriorating.
* Histological or cytological proof of adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.
* Presence of a pathogenic homologous recombination repair mutation in at least one of the following genes on tumor tissue or circulating tumor DNA testing: BRCA1, BRCA2, ATM (limited to 15% of enrolled participants), CDK12, CHEK2, PALB2, MLH1, NBN, ATR, FANCA, MRE11A, RAD51C. Assessment of HRR mutation status by germline or somatic testing. All testing must be per Clinical Laboratory Improvement Amendments (CLIA)-certified assay and may have occurred at any time prior to or at screening (not required to be completed within the screening window).
* Metastatic castration-resistant prostate cancer (mCRPC) as demonstrated by one of the following:

  * Metastatic disease documented by conventional imaging: computed tomography (CT)/magnetic resonance imaging (MRI) chest/abdomen/pelvis and bone scan are required to be performed, but metastases do not need to be seen on both modalities. Measurable disease is not required.
  * Unequivocal prostate-specific membrane antigen (PSMA) positron emission tomography (PET) only defined metastatic disease with negative conventional imaging. PSMA PET imaging is not required to be performed, but may be used to document metastases when relevant.
* Received prior abiraterone acetate with prednisone for mHSPC or locally advanced disease and on which progressed via a minimum of 2 rising PSA levels with a minimum of a 1-week interval between each determination or radiographic progression by any form of imaging.
* Progressive disease at start of treatment and in the setting of medical or surgical castration as defined by 1 or more of the following 4 criteria:

  * PSA progression defined as 2 rising PSA levels, above an initial reference value, taken with a minimum of a 1-week interval. If PSA rise is the only indication of progression at start of study treatment, a minimum PSA of 1.0 ng/mL is required and all measured PSA values have to be considered to make a determination of progression.
  * Soft tissue disease progression as defined by RECIST 1.1.
  * Bone disease progression defined by PCWG3 with 2 or more new metastatic bone lesions on a whole-body radionuclide bone scan.
  * Appearance of newly identified, convincingly positive lesions consistent with metastatic prostate cancer on PSMA PET.
* Surgically or medically castrated, with testosterone levels of <50 ng/dL. If the participant is medically castrated, continuous dosing with a gonadotropin-releasing hormone agonist or antagonist must be demonstrated by testosterone level of <50 ng/dL and planned to continue throughout study participation.
* Eastern Cooperative Oncology Group (ECOG) status of ≤1 (Appendix A: Performance Status Criteria).
* Normal organ function with acceptable initial laboratory values within 14 days of treatment start:

  * Absolute neutrophil count ≥ 1,500/µl
  * Hemoglobin ≥ 9g/dl
  * Platelet count ≥ 100,000/µl
  * Creatinine ≤ 1.5 x the institutional upper limit of normal (ULN)
  * Potassium ≥ 3.5 mmol/L (within institutional normal range)
  * Bilirubin ≤ 1.3 x ULN (unless documented Gilbert's disease)
  * Serum glutamic oxaloacetic transaminase/aspartate transaminase (AST) ≤ 2.5 x ULN
  * Serum glutamic pyruvic transaminase/ alanine transaminase (ALT) ≤ 2.5 x ULN
* Participants must agree to use a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including 4 months after the last dose of study drug. Sperm donation is prohibited during the study and for 4 months after the last dose of study drug. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.

Exclusion Criteria

* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer or superficial bladder cancer.
* Prior treatment for metastatic or non-metastatic CRPC with an ARPI other than abiraterone acetate with prednisone for ≥ 12 weeks. Prior treatment with abiraterone acetate with prednisone in the mHSPC or locally advanced setting is not exclusionary.
* Participants who received chemotherapy for castration-sensitive prostate cancer are still eligible provided chemotherapy was completed >6 months prior to start of study treatment.
* Use of investigational agents for the treatment of prostate cancer within 4 weeks of start of study treatment.
* Prior treatment with a PARP inhibitor.
* Concurrent treatment with crizotinib.
* Prior platinum-based chemotherapy for the treatment of prostate cancer.
* Current or planned use of potent P-gp inhibitors within 7 days prior to randomization. The P-gp inhibitors include: amiodarone, carvedilol, clarithromycin, cobicistat, dronedarone, erythromycin, glecaprevir/pibrentasvir, indinavir, itraconazole, ketoconazole, lapatinib, lopinavir, propafenone, quinidine, ranolazine, ritonavir, saquinavir, sofosbuvir/velpatasvir/voxilaprevir, telaprevir, tipranavir, valspodar, and verapamil.
* Current use of strong cytochrome P450 2C8 (CYP2C8) inhibitors (e.g., clopidogrel, gemfibrozil) and inducers (e.g., rifampin), strong CYP3A4 inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine and St. John's Wort), moderate CYP3A4 inducers (e.g., bosentan, efavirenz, etravirine, modafinil and nafcillin), or substrates of CYP3A4 (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus and tacrolimus), CYP2C9 (e.g., phenytoin, warfarin), or CYP2C19 (e.g., S-mephenytoin) with a narrow therapeutic index unless considered medically necessary to treat a life-threatening condition.
* Participants treated with strong cytochrome P450 2C8 (CYP2C8) inhibitors (e.g., clopidogrel, gemfibrozil) within 7 days from randomization are not eligible.
* Use of hormonal agents with anti-tumor activity against prostate cancer including 5-alpha reductase inhibitors, androgens (e.g., testosterone), cytoproterone acetate, progestational agents, and estrogens/diethylstilbestrol within 28 days prior to the start of study treatment.
* Use of herbal products or alternative therapies that may decrease PSA levels or that may have hormonal anti-prostate cancer activity (e.g., saw palmetto, PC-SPES, PC-HOPE, St. John's wort, selenium supplements, grape seed extract, etc.) within 28 days of study treatment initiation or plans to initiate treatment with these products/alternative therapies during the entire duration of the study.
* Participants receiving a blood transfusion within 14 days of randomization are not eligible.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma). Also, history of loss of consciousness or transient ischemic attack within 12 months of randomization.
* Medical conditions such as uncontrolled hypertension as indicated by a resting systolic blood pressure > 160 mm Hg or diastolic blood pressure > 90 mm Hg at screening, uncontrolled diabetes mellitus, and cardiac disease that would preclude participation, as determined by the investigator.
* Untreated known or suspected brain metastases or spinal cord compression or clinically significant malignant epidural disease.
* Use of any prohibited concomitant medications (Appendix C: Medications with the Potential for Drug-Drug Interactions) within 28 days before first dose of study treatment.
* Grade >2 treatment-related toxicity from prior therapy except alopecia or peripheral neuropathy.
* Known allergy to any of the compounds under investigation.
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
radiographic progression free survival (rPFS) | From treatment initiation until documented disease progression, death, lost to follow-up, withdrawal, administrative censoring at the time of final analysis, assessed at approximately 42 months from the start of enrollment.
  To compare the efficacy of talazoparib + enzalutamide to talazoparib alone as measured by rPFS as assessed by the Investigator.

SECONDARY OUTCOMES:
Time to PSA50 | Time from treatment initiation until observed PSA50, assessed at approximately 42 months from the start of enrollment.
  To compare the efficacy of talazoparib + enzalutamide to talazoparib alone as measured by time to prostate specific antigen (PSA) ≥ 50% decline.
Time to PSA Progression | From treatment initiation until documented PSA progression, assessed at approximately 42 months from the start of enrollment.
  To compare the efficacy of talazoparib + enzalutamide to talazoparib alone as measured by time to PSA progression.
Quality of Life (QoL) by Functional Assessment of Cancer Therapy-Prostate (FACT-P) | From prior to treatment initiation (screening) until treatment discontinuation, assessed at approximately 42 months from the start of enrollment.
  Overall QoL measured by FACT-P. Scales: FACT-P Total score (range 0-156), FACT-General (G) Total score (range 0-108), FACT-P Trial Outcome Index (TOI) score (range 0-104). The higher the score, the better the QOL.
Quality of Life (QoL) by Functional Assessment of Cancer Intervention Therapy-Fatigue Scale (FACIT-Fatigue) | From prior to treatment initiation (screening) until treatment discontinuation, assessed at approximately 42 months from the start of enrollment.
  Fatigue measured by FACIT-Fatigue. Scales: FACIT-F Total score (range 0-160), FACT-General (G) Total score (range 0-108), FACIT-F Trial Outcome Index (TOI) score (range 0-108). The higher the score, the better the QOL.
Quality of Life (QoL) by Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | From prior to treatment initiation (screening) until treatment discontinuation, assessed at approximately 42 months from the start of enrollment.
  Cognitive function measured by FACT-Cog. Subscales: Perceived Cognitive Impairments (CogPCI) score (range 0-72), Impact of Perceived Cognitive Impairments on Quality of Life (CogQOL) score (range 0-16), Comments from Others (CogOth) score (range 0-16), Perceived Cognitive Abilities (CogPCA) score (range 0-28). The higher the score, the better the QOL.
Adverse Events (AE) | From treatment initiation through follow up, up to 12 months from end of treatment, assessed at approximately 42 months from the start of enrollment.
  Evaluate AE occurrence according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 to confirm safety.
Overall Survival (OS) | From treatment initiation until death, lost to follow-up, withdrawal, administrative censoring at the time of final analysis, assessed at approximately 42 months from the start of enrollment.
  To compare the efficacy of talazoparib + enzalutamide to talazoparib alone as measured by OS.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Morgans, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Prostate Cancer Clinical Trials Consortium, LLC supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: pcctc@mskcc.org.
Supporting Information: ICF